CLINICAL TRIAL: NCT00770627
Title: A Randomized , Controlled, Doulbe Blind Placebo Trial To Evaluate The Efficacy and the Tolerance of an Omega 3 Fatty Acids Supplementation in ADHD Children
Brief Title: Clinical Trial to Evaluate the Efficacy and the Tolerance of an Omega 3 Fatty Acids Supplementation in ADHD Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Doctor Olivier Revol, Pierre Wertheimer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F-08-08-3103039
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: 160 children; parallel group
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo caps (Placebo Comparator)
  Interventions: Dietary Supplement: Omega 3 caps
- Omega 3 caps (Active Comparator)
  Interventions: Dietary Supplement: Omega 3 caps

INTERVENTIONS:
Dietary Supplement: Omega 3 caps — Children between 6 and 8 years must take 2 caps/day Children between 9 and 11 years must take 3 caps/day Children between 12 and 15 years must take 4 caps /day

SUMMARY:
Principal focus is to evaluate the effects of omega 3 fatty acids supplementation on the ADHD children's behaviour during 12 weeks on two years. The secondary focus is to evaluate the effects of omega 3 fatty acids supplementation on the lexical level,intentional abilities, anxiety and depression.

The omega 3 fatty acids don't present adverse side effects. The inclusion to the trial could avoid the intake the methylphenidate and its associated adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 15 years and 11 months of age ADHD children with hyperactivity confirmed dy DSM IV criteria Children and parents' consent

Exclusion Criteria:

* Without methylphenidate treatment Fish or other sea products allergic Intake of sea omega 3 fatty acids supplments more one week during 3 months before the trial Children need quickly to take methylphenidate: social, family, or school risk Intake methylphenidate 30 days before the trial or/and intake it during one consecutive week

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
ADHD rating scale | 5 minutes

SECONDARY OUTCOMES:
Conners (parents, 48 items), CDI (Depression), Tête de l'alouette (lexical capacity), KITAP Battery (Attentional capacity) | 3 hours

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinical Investigation Center, Bron
  - Hopital Cardiovasculaire Louis Pradel, Bron

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600